CLINICAL TRIAL: NCT01367743
Title: Optimizing the Use of Vasopressor After Coronary Reperfusion in Cardiogenic Shock Secondary to Myocardial Infarction. Pathophysiological Study Comparing the Efficacy and Cardio-circulatory Tolerability of Epinephrine and Norepinephrine
Brief Title: Study Comparing the Efficacy and Tolerability of Epinephrine and Norepinephrine in Cardiogenic Shock
Acronym: OptimaCC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-017081-23
Record Dates: First submitted 2011-05-10; First posted 2011-06-07 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Cardiogenic Shock
Keywords: myocardial infarction; epinephrine; norepinephrine; cardiac output
MeSH Terms: conditions — Shock, Cardiogenic; Myocardial Infarction | interventions — Vasoconstrictor Agents; Catecholamines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- epinephrine (Active Comparator)
  Interventions: Drug: epinephrine perfusion
- norepinephrine (Active Comparator)
  Interventions: Drug: norepinephrine perfusion

INTERVENTIONS:
Drug: epinephrine perfusion — perfusion of commercial epinephrine prepared in syringes in order to obtain a MAP of 65-70 mmHg
  Other Names: vasopressor; catecholamine
  Arms: epinephrine
Drug: norepinephrine perfusion — perfusion of commercial norepinephrine prepared in syringes in order to obtain a MAP of 65-70 mmHg
  Other Names: vasopressor; catecholamine
  Arms: norepinephrine

SUMMARY:
The efficacy and tolerability of norepinephrine and epinephrine in cardiogenic shock after reperfused myocardial infarction will be compared, by following cardiac index evolution as main criteria. The study is a pilot pathophysiological study, randomized, double blind and multicenter.

DETAILED DESCRIPTION:
Cardiogenic shock secondary to myocardial infarction is a frequent pathology in reanimation and is associated with high mortality (50%). Hemodynamic management and notably the choice of vasopressor in cardiogenic shock states secondary to myocardial infarction (cardiac index < 2.2 l/min/m-2) is not codified. There are two opposite views: a) the first is based on the fact that an hypotensive patient with low cardiac output is primarily in need of an inotropic agent and that, consequently, epinephrine is the molecule of choice (inotropic and vasoconstrictor); b) the second is based on the fact that hypotension also reflects a certain degree of vascular failure and vascular vasoplegia and therefore norepinephrine is the molecule of choice along with, if needed, the eventual addition of dobutamine in order to separately titrate vasoconstriction and inotropism.

Study hypotheses: epinephrine could facilitate myocardial function by providing the latter with its preferred substrate (lactate) and thus induce a higher cardiac index along with increased energy expenditure. Norepinephrine is the therapy of choice of hypotensive states; nevertheless its lack of inotropic effect could theoretically exacerbate myocardial failure. Thus, the aim of the study is to compared the efficiency and the tolerability of norepinephrine and epinephrine in cardiogenic shock after reperfused myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* man or woman older than 18 years
* cardiogenic shock due to myocardial infarction treated by angioplasty
* SAP < 90 MM Hg or MAP < 65 mm Hg without vasopressor or vasopressor necessity
* sign of tissue hypoperfusion
* cardiac index < 2.2 l/mn/m2 in the absence of vasopressive or inotropic therapy
* pulmonary artery occlusion pressure > 15 mmHg or echocardiographic evidence of high pressure (mitral profile)
* exclusion of covert hypovolemia : Delta PP if feasible should be > 13% (patient adapted to the ventilator and sinus rhythm) and /or no response to passive leg raising
* ejection fraction < 40% in ultrasound without inotrope support. This criteria will not be taken into account in instances of treatment with dopamine, norepinephrine, epinephrine, dobutamine or milrinone.

Exclusion Criteria:

* shock of other origin
* immediate indications for mechanical assistance device
* minor aged patients
* patients for whom written consent - by patient or family - has not been obtained. Given the seriousness of the medical situation at the time of inclusion, patient consent will be difficult if not impossible to obtain. The inclusion will only be possible after information is provided and consent is obtained from a family member. As soon as possible, protocol information will be issued to the patient in order to obtain consent for continuance.
* cardiac arrest with early signs of cerebral anoxia.
* septic, toxic and obstructive cardiomyopathy
* arrhythmogenic cardiomyopathy
* patient with coronary insufficiency
* patient with ventricular rhythm disorders
* patient treated with a medicine listed in contre indication
* patient without social assurance
* patient major under legal protection or safeguard justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-09; Primary Completion 2016-02 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Compared effects of investigated drugs on cardiac index | H0; H2, H4, H6, H12, H24, H48 and H72
  effectiveness of the treatment assessed by the evolution of cardiac index

SECONDARY OUTCOMES:
pro/anti-inflammatory cytokines | H0, H24, H48 and H72
  Compared effects of investigated drugs on pro/anti-inflammatory cytokines
BNP | H0, H24, H48 and H72
  Compared effects of investigated drugs on BNP
Troponin | H0, H24, H48 and H72
  Compared effects of investigated drugs on Troponin
catecholamine doses | H0, H24, H48 and H72
  Compared effects of investigated drugs on the catecholamine doses
organ failure (SOFA Score) | H0, H24, H48 and H72
  Compared effects of investigated drugs on the organ failure
Lactate clearance | H0, H2, H6, H12, H24 and H48
  Compared effects of investigated drugs on the Lactate clearance
heart rate | H0, H2, H4, H6, H12, H24, H48 and H72
  Compared effects of investigated drugs on heart rate and the incidence of arrhythmia
cardiac power index | H0, H2, H4, H6, H12, H24, H48 and H72.
  Compared effects of investigated drugs on cardiac power
SVO2 | H0, H2, H4, H6, H12, H24, H48 and H72.
  Compared effects of investigated drugs on the SVO2
cardiac double product | H0, H2, H4, H6, H12, H24, H48 and H72.
  Compared effects of investigated drugs on the cardiac double product
refractory cardiogenic shock | H0, H2, H4, H6, H12, H24, H48 and H72.
  compared effects of the investigated drugs on the occurrence of refractory cardiogenic shock

CONTACTS AND LOCATIONS:
Overall Officials: Philippe VIGNON, Dr, Principal Investigator — CHU Limoges
Locations (11):
- France (11):
  - Nancy Brabois university hospital, Vandœuvre-lès-Nancy, Meurthe Et Moselle
  - CHU de BESANCON / Hôpital Jean Minjoz, Besançon
  - CHU de DIJON, Dijon
  - CHU de LIMOGES Hôpital Dupuytren, Limoges
  - APHM Hôpital NORD, Marseille
  - Chr Metz Thionville, Metz
  - CH de MULHOUSE, Mulhouse
  - AP-HP-Hôpital Cochin, Paris
  - CHU de STRASBOURG / NHC, Strasbourg
  - CHU Toulouse, Toulouse
  - Chru Tours, Tours

REFERENCES:
- [Derived] Takagi K, Blet A, Levy B, Deniau B, Azibani F, Feliot E, Bergmann A, Santos K, Hartmann O, Gayat E, Mebazaa A, Kimmoun A. Circulating dipeptidyl peptidase 3 and alteration in haemodynamics in cardiogenic shock: results from the OptimaCC trial. Eur J Heart Fail. 2020 Feb;22(2):279-286. doi: 10.1002/ejhf.1600. Epub 2019 Aug 31. PMID 31472039
- [Derived] Levy B, Clere-Jehl R, Legras A, Morichau-Beauchant T, Leone M, Frederique G, Quenot JP, Kimmoun A, Cariou A, Lassus J, Harjola VP, Meziani F, Louis G, Rossignol P, Duarte K, Girerd N, Mebazaa A, Vignon P; Collaborators. Epinephrine Versus Norepinephrine for Cardiogenic Shock After Acute Myocardial Infarction. J Am Coll Cardiol. 2018 Jul 10;72(2):173-182. doi: 10.1016/j.jacc.2018.04.051. PMID 29976291
- Available data/document: Statistical Analysis Plan — http://cic-p-nancy.fr/wp-content/uploads/2019/01/revUS_SAP_OPTIMA_CC_KD_NG.pdf